CLINICAL TRIAL: NCT03852862
Title: Double Regional Anesthesia in Video Assisted Thoracoscopy
Acronym: DRAVATS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/182/HP
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Video Assisted Thoracoscopy; Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus plane block with paravertebral block (Experimental): Association of Serratus plane block and paravertebral block for anesthesia
  Interventions: Drug: Serratus plane block and paravertebral block
- paravertebral block alone (Active Comparator): Paravertebral block for anesthesia
  Interventions: Drug: paravertebral block

INTERVENTIONS:
Drug: Serratus plane block and paravertebral block — Single Administration of 20 mL of ropivacaine for Serratus plane block (Intra-muscular injection) followed by a single administration of 20 ml ropivacaine for paravertebral block (T4 inter-vertebral injection)
  Arms: Serratus plane block with paravertebral block
Drug: paravertebral block — Single Administration of 20 ml of ropivacaine for paravertebral block (T4 inter-vertebral injection)
  Arms: paravertebral block alone

SUMMARY:
Monocentric, randomized, controlled, single-blind study who's aim is to demonstrate the efficacy of the association of paravertebral block and serratus plane block with paravertebral block alone

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 75 years;
* Programmed for unilateral videothoracoscopy for anatomical resection (segmentectomy, lobectomy);
* Subject affiliated to a social security scheme;
* Subject having signed an informed consent

Exclusion Criteria:

* Chronic treatment with opiates;
* Contraindication to administration of morphine;
* Allergy to local anesthetics or contraindications to the use of ropivacaine;
* Contraindication to the realization of paravertebral blocks and serratus;
* Pregnancy, breastfeeding;
* Severe obesity (BMI > 40 kg/m²);
* Renal impairment (GFR < 30 mL/min) or known severe hepatic impairment;
* Difficulties of comprehension preventing the collection of consent and the realization of the study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Number of opioids drug administrated | 24 hours postoperatively

SECONDARY OUTCOMES:
Length of stay in recovery room | 24 hours postoperatively
Total duration of hospitalization | during the 28 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Melody DUSSEAUX, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France